CLINICAL TRIAL: NCT05423392
Title: Efficacy of 4% Articaine Terminal Anesthesia in the Lateral Jaw Region in Children: A Double-blind Randomized Study
Brief Title: Efficacy of 4% Articaine Terminal Anesthesia in the Lateral Jaw Region in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Branislav Bajkin, MD, DMD, PhD, Full Professor, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-18/12-2020
Record Dates: First submitted 2022-01-11; First posted 2022-06-21 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Dental Caries; Primary Teeth; Inferior Alveolar Nerve; Anesthesia, Dental
Keywords: Carticaine; Anesthesia, Dental; Pediatric Dentistry
MeSH Terms: conditions — Dental Caries | interventions — Carticaine

STUDY DESIGN:
Intervention Model Description: A RANDOMIZED DOUBLE BLIND
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomly and equally assigned to treatment groups. The study was planned as a double-blind. Thus, neither the patients nor the researchers knew which anesthetic will be applied. Only practioner, who will injected anesthetic will know what tipe of anesthetic is it - 4% articain or 2% lidocain chlorid. Number of participials is 60, divided into two equal groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The first tasted group using 4% Articaine (Experimental): The group was divided into three subgroups depending on the age of the participials: 1st group from 5-9 years, 2nd from 10-13 years and 3th from 14-18 years.
  Following placement of 5% lidocaine topical anaesthetic for 3 minutes prior to and at the site of needle penetration, patients were randomly given one of the following local anesthetic regimes administered by the principle investigator. For indicated dental treatment patients would receive 2.0 ml 4% articaine with 1:100,000 epinephrine as a local infiltration in the mucobuccal region,the lateral region of the lower jaw.Criteria for measuring efficacy would be to measure pain during anesthetic injection, 10 minutes after injection,during and after the intervention. The child's behavior would be monitored through all phases of clinical work by direct observation of the dentist( examiner) using the above methodology. After that, the examiner would fill in the questionnaire based on the answer of the child / parent (guardian).
  Interventions: Procedure: Tooth extraction of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years; Procedure: Endodontic dental treatment of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years; Procedure: Conservative tooth restoration of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years
- The second tasted group using 2% Lidocaine-chloride (Active Comparator): The group was divided into three subgroups depending on the age of the participials: 1st group from 5-9 years, 2nd from 10-13 years and 3th from 14-18 years. Following placement of 5% lidocaine topical anesthetic for 3 minutes prior to and at the site of needle penetration, patients were randomly given one of the following local anesthetic regimes administered by the principle investigator. For the indicated dental treatment will be used 2.0 ml 2% lidocaine with 1:80,000 epinephrine as an IANB anesthesia for n.alveolaris inferior. Criteria for measuring efficacy would be to measure pain during anesthetic injection, 10 minutes after injection,during and after the intervention. The child's behavior would be monitored through all phases of clinical work by direct observation of the dentist( examiner) using the above methodology. After that, the examiner would fill in the questionnaire based on the answer of the child / parent (guardian).
  Interventions: Procedure: Tooth extraction of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years; Procedure: Endodontic dental treatment of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years; Procedure: Conservative tooth restoration of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years

INTERVENTIONS:
Procedure: Tooth extraction of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years — Tooth extraction will be following up with the methodological procedures in order to define the effectiveness of anesthetics during indicated dental procedure.
  Other Names: 4% Articaine; Effectiveness of anesthetics; Lateral jaw region in children; 2% Lidocaine-chloride
Procedure: Endodontic dental treatment of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years — Endodontic dental treatment will be following up with the methodological procedures in order to define the effectiveness of anesthetics during dental treatment.
  Other Names: 4% Articaine; Effectiveness of anesthetics; Lateral jaw region in children; 2% Lidocaine-chloride
Procedure: Conservative tooth restoration of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years — Conservative tooth restoration will be following up with the methodological procedures in order to define the effectiveness of anesthetics during conservative tooth restoration.
  Other Names: 4% Articaine; Effectiveness of anesthetics; Lateral jaw region in children; 2% Lidocaine-chloride

SUMMARY:
Optimal anesthesia is an essential requirement for successful dentoalveolar intervention.To achieve this goal,different anesthetic agents and techniques are available. Inferior alveolar nerve block (IANB) remains the most commonly used anesthetic technique. However, after the worldwide approval of articaine, a relatively new local anesthetic with enhanced tissue diffusion properties, many studies on healthy volunteers have investigated the anesthetic efficacy of buccal articaine infiltration and IANB in the mandibular posterior teeth and reported comparable results. Infiltration anesthesia is technically more straightforward, less stressful to the patient, and associated with higher success and lower complication rates than block anesthesia. The aim of this study was to determine the effectiveness of local infiltration anesthesia using 4% articaine in the analgesia of deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years.

DETAILED DESCRIPTION:
Clinical study to evaluate the effectiveness of local anesthesia with 4% articaine in order to ensure painless and effective implementation of dental procedures in children. Selection of respondents: participians with good systemic health - patients classified as American Society of Anesthesiologists (ASA) classification - ASA I and ASA II will be included in the study and required invasive dental treatment using local anesthetic (restoration or extraction) on deciduous and permanent molars in children aged 5-18 years and mandibular premolars in children aged 10-18 years, over 20 kg of body weight.The research would include at least 60 participials aged 5-18, who would be divided into two groups. One group the local anesthetic 4% articaine would be used. The second group would be provided with the local anesthetic 2% lidocaine chloride, as a control group. Analysis and data collection in each group would create subgroups depending on the age of the participials: 5-9 years, 10-13 years and 14-18 years.A clinical study would be doubly blind. Participials who would be included in the clinical study would sign a consent form to participate in the clinical study but would not know which anesthetic would be received.Criteria for measuring efficacy would be to measure pain during anesthetic injection,10 minutes after injection, and during and after the intervention using:

1. Visual Analog Scales (VAS)
2. Tooth vitality test
3. Wong-Baker Pain Rating Scale (W-BFSR)
4. Frank Behavior Rating Scale (FBRS)
5. By determining the growth and development of the roots of permanent premolars and molars
6. By determining the resorption of the roots of deciduous molars.

The child's behavior would be monitored through all phases of clinical work by direct observation of the dentist(examiner) who is in charge of measuring the effectiveness of anesthetics but does not know what type of anesthetic. Only a dentist who applies(practitioner) an anesthetic will know what type of anesthetic it is. After that, the examiner would fill in the questionnaire based on the answer of the child / parent (guardian).

In accordance with known ethical principles and in accordance with the principles of Good Clinical Practice (GCP), care for the well-being of the patients was maximally respected, in accordance with the latest revision of the Declaration of Helsinki and accepted principles that apply to clinical trials on humans. The holder of the protection of the patients in this clinical trial is the principal researcher, who cooperated with the Ethics Committee of the Dental Clinic of Vojvodina, University of Novi Sad. The patients written Informed Consent implied that the patient had received full information about the research, and was stressed that they had the right to decide independently to participate, without coercion and external influences, or any harmful consequences if they refused to participate.

ELIGIBILITY:
Inclusion Criteria:

* Respondents of both sexes, aged 5-18 years
* Subjects in need of either conservative rehabilitation or tooth extraction on deciduous or permanent premolars and / or molars
* Subjects who have an X-ray of the teeth for the need of dental rehabilitation

Exclusion Criteria:

* difficult cooperation with the patient
* existence of allergy to local anesthetic
* the existence of a diagnosed general disease
* unsigned informative consent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Checkout of painlessness in lateral region lower jaw in children using Visual Analog Scale | during procedure
  Checkout of painlessness in lateral region lower jaw in children using Visual Analog Scale from 0 to 10, where 0 means absence of pain and 10 means unbearable pain.
Checkout of painlessness in lateral region lower jaw in children using tooth vitality test | 10 minutes after anesthetic injection
  Control and verification of painlessness of the anesthetized lower jaw region will be performed 10 minutes after anesthetic injection using a tooth vitality test.
Checkout of painlessness in lateral region lower jaw in children using Wong-Baker Pain Rating Scale | during procedure
  Checkout of painlessness in lateral region lower jaw in children using Wong-Baker Pain Rating Scale from 0 to 10, where 0 means absence of pain and 10 means the strongest possible pain.
Checkout of painlessness in lateral region lower jaw in children using Frank Behavior Rating Scale | during procedure
  Checkout of painlessness in lateral region lower jaw in children using Frank Behavior Rating Scale from 0 to 2 , where 0 means cooperating patient and 2 means complete lack of cooperation.
Checkout of painlessness in lateral region lower jaw in children by determining the development of the roots of permanent teeth | before intervention
  By determining the growth and development of the roots of permanent premolars and molars by examiner using x-ray before intervention.
Checkout of painlessness in lateral region lower jaw in children by determining the resorption of the roots of deciduous teeth | before intervention
  By determining the resorption of the roots of deciduous molars by examiner using x-ray before intervention.

SECONDARY OUTCOMES:
Success of indicated dental treatment using tooth vitality test | 10 minutes after dental treatment
  The success and effectiveness of anesthetics will be determined immediately after the completion of the indicated dental treatment using tooth vitality test 10 minutes after dental treatment.
Success of indicated dental treatment using Visual Analog Scale | immediately after dental treatment
  The success and effectiveness of anesthetics will be determined immediately after the completion of the indicated dental treatment using Visual Analog Scale from 0 to 10, where 0 means absence of pain and 10 means unbearable pain.
Success of indicated dental treatment using Wong-Baker Pain Rating Scale | immediately after dental treatment
  The success and effectiveness of anesthetics will be determined immediately after the completion of the indicated dental treatment using Wong-Baker Pain Rating Scale from 0 to 10, where 0 means absence of pain and 10 means the strongest possible pain.
Success of indicated dental treatment using Frank Behavior Rating Scale | immediately after dental treatment
  The success and effectiveness of anesthetics will be determined immediately after the completion of the indicated dental treatment using Frank Behavior Rating Scale from 0 to 2 , where 0 means cooperating patient and 2 means complete lack of cooperation.

OTHER OUTCOMES:
Success of indicated dental treatment using questionnaire | 15 minutes after dental treatment
  The examiner would fill in a questionnaire ( The guestionnaire for the child / parent (guardian)) wich contains 10 questions with YES or NO answers about the dental procedure and the success of the indicated treatment based on children's responses. Five and more positive answers of ten questions support the positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Branislav V Bajkin, DMD, PhD, Study Chair — Dental Clinic of Vojvodina, Faculty of Medicine, University of Novi Sad; Jelena Komšić, DMD, Study Director — Dental Clinic of Vojvodina, Faculty of Medicine, University of Novi Sad
Locations (1):
- Dental Clinic of Vojvodina, Faculty of Medicine, University of Novi Sad, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Majid OW, Ahmed AM. The Anesthetic Efficacy of Articaine and Lidocaine in Equivalent Doses as Buccal and Non-Palatal Infiltration for Maxillary Molar Extraction: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial. J Oral Maxillofac Surg. 2018 Apr;76(4):737-743. doi: 10.1016/j.joms.2017.11.028. Epub 2017 Nov 27. PMID 29257943
- [Result] Malamed SF, Handbook of Local Anaesthesia, 4th ed. St. Louis: Mosby-Year Book; 1997. pp. 63-64.
- [Result] Peedikayil FC, Vijayan A. An update on local anesthesia for pediatric dental patients. Anesth Essays Res. 2013 Jan-Apr;7(1):4-9. doi: 10.4103/0259-1162.113977. PMID 25885712
- [Result] Alzahrani F, Duggal MS, Munyombwe T, Tahmassebi JF. Anaesthetic efficacy of 4% articaine and 2% lidocaine for extraction and pulpotomy of mandibular primary molars: an equivalence parallel prospective randomized controlled trial. Int J Paediatr Dent. 2018 May;28(3):335-344. doi: 10.1111/ipd.12361. Epub 2018 Mar 24. PMID 29573375
- [Result] Arrow P. A comparison of articaine 4% and lignocaine 2% in block and infiltration analgesia in children. Aust Dent J. 2012 Sep;57(3):325-33. doi: 10.1111/j.1834-7819.2012.01699.x. Epub 2012 May 28. PMID 22924356
- [Result] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Result] Hockenberry MJ, Wilson D, Winkelstein ML. Wongs Essentials of Pediatric Nursing. 7th end. St Louis: Mosby, 2005: 1259.
- [Result] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Result] Champion GD, Goodenough B, von Baeyer CL, Thomas W. Measurement of Pain in Infants and Children, Progress in Pain Research and Management , vol 10. Seattle: IASP Press, 1998: 123-160.
- [Result] Meechan JG. The use of the mandibular infiltration anesthetic technique in adults. J Am Dent Assoc. 2011 Sep;142 Suppl 3:19S-24S. doi: 10.14219/jada.archive.2011.0343. PMID 21881058
- [Result] Oulis CJ, Vadiakas GP, Vasilopoulou A. The effectiveness of mandibular infiltration compared to mandibular block anesthesia in treating primary molars in children. Pediatr Dent. 1996 Jul-Aug;18(4):301-5. PMID 8857658
- [Result] Jung IY, Kim JH, Kim ES, Lee CY, Lee SJ. An evaluation of buccal infiltrations and inferior alveolar nerve blocks in pulpal anesthesia for mandibular first molars. J Endod. 2008 Jan;34(1):11-3. doi: 10.1016/j.joen.2007.09.006. PMID 18155484
- [Result] Corbett IP, Kanaa MD, Whitworth JM, Meechan JG. Articaine infiltration for anesthesia of mandibular first molars. J Endod. 2008 May;34(5):514-8. doi: 10.1016/j.joen.2008.02.042. PMID 18436027
- [Result] Srinivasan MR, Poorni S, Nitharshika Y, et al: Articaine buccal infiltration versus lignocaine inferior alveolar block for pulpal anesthesia in mandibular second premolars-Randomized control double blinded clinical trial. J Pierre Fauchard Acad 31:79, 2017
- [Result] Meechan JG. Infiltration anesthesia in the mandible. Dent Clin North Am. 2010 Oct;54(4):621-9. doi: 10.1016/j.cden.2010.06.003. PMID 20831926